CLINICAL TRIAL: NCT00401973
Title: The Assessment of the Safety, Efficacy, and Practicality of an Algorithm Including Amantadine, Metformin and Zonisamide for the Prevention of Olanzapine-Associated Weight Gain in Outpatients With Schizophrenia
Brief Title: Assessment of Safety and Efficacy of Therapy for the Prevention of Weight Gain Associated With Olanzapine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10768; F1D-US-HGMM
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2009-09-30 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-09

CONDITIONS: Schizophrenia; Schizoaffective Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine; Amantadine; Metformin; Zonisamide

ARMS (3):
- Olanzapine (Experimental): olanzapine plus behavioral information
  Interventions: Drug: olanzapine; Behavioral: Wellness education
- Olanzapine + Amantadine (Experimental): Olanzapine and Pharmacological Algorithm 1a - amantadine first plus behavioral information
  Interventions: Drug: olanzapine; Drug: amantadine; Drug: metformin; Drug: zonisamide; Behavioral: Wellness education
- Olanzapine + Metformin (Experimental): Olanzapine and Pharmacological Algorithm 1b - metformin first plus behavioral information
  Interventions: Drug: olanzapine; Drug: amantadine; Drug: metformin; Drug: zonisamide; Behavioral: Wellness education

INTERVENTIONS:
Drug: olanzapine — 5-20 milligrams (mg), oral, daily for 22 weeks.
  Other Names: LY170053; Zyprexa
Drug: amantadine — Amantadine, 100 milligrams (mg), oral, 1 twice a day (BID). Patients who gained greater than 3 kilograms (kg) will switch to metformin. Patients who gained greater than 3 kg after switching to metformin will be switched to zonisamide.
  Arms: Olanzapine + Amantadine; Olanzapine + Metformin
Drug: metformin — Metformin, 500 mg, oral, twice a day (BID) for 2 weeks titrated to 500mg three times a day (TID) thereafter. Patients who gain greater than 3 kilograms (kg) will be switched to amantadine. Patients who gained greater than 3 kg after switching to amantadine will be switched to zonisamide.
  Arms: Olanzapine + Amantadine; Olanzapine + Metformin
Drug: zonisamide — Zonisamide, 100-400mg, oral, daily.
  Arms: Olanzapine + Amantadine; Olanzapine + Metformin
Behavioral: Wellness education — weight management

SUMMARY:
The goal of this study is to answer the following questions:

* Whether treatment with amantadine, metformin or zonisamide can prevent or reverse the weight gain that is associated with olanzapine
* Whether taking amantadine, metformin or zonisamide can help patients decrease or eliminate some of the changes in body that occur with weight gain
* How weight gain associated with olanzapine can affect people
* Whether treatment with amantadine, metformin or zonisamide can help eliminate weight gain associated with olanzapine and not interfere with the positive effects of olanzapine on functioning of people with schizophrenia and other diseases

ELIGIBILITY:
Inclusion Criteria:

* You must have been diagnosed with schizophrenia or schizoaffective disorder
* You must be able to visit the doctor's office once every two weeks for three months, then once every four weeks for the next three months with a possible bi-weekly visit during the fifth month
* If you are currently taking a medication for schizophrenia or schizoaffective disorder, you have been taking it for at least 30 days without any changes
* If you are a female, you must have a negative pregnancy test and be using an effective method of contraception

Exclusion Criteria:

* You have a diagnosis of bipolar I disorder, diabetes, very high triglyceride level (fasting triglycerides greater than or equal to 500 mg/dL), recent heart attack, stroke, uncontrolled seizures, serious infection, unstable heart disease (such as ischemic heart disease or congestive heart failure), an uncorrected narrow angle glaucoma or human immunodeficiency virus (HIV)
* You have diseases of the intestinal tract, lungs, liver, kidney, nervous or endocrine systems, or blood
* You have a diagnosis of an eating disorder
* You have a history of Parkinson's Disease or any related disorders
* You are allergic to sulfa drugs or any of the medications involved in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Canton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnson City, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeSoto, Texas
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rio de Janeiro
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salvador
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beer Yaacov, Israel
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City, Mexico
- Puerto Rico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bayamón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow, Russia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul, South Korea

REFERENCES:
- [Derived] Hoffmann VP, Case M, Jacobson JG. Assessment of treatment algorithms including amantadine, metformin, and zonisamide for the prevention of weight gain with olanzapine: a randomized controlled open-label study. J Clin Psychiatry. 2012 Feb;73(2):216-23. doi: 10.4088/JCP.09m05580. Epub 2011 May 17. PMID 21672497
- [Derived] Case M, Treuer T, Karagianis J, Hoffmann VP. The potential role of appetite in predicting weight changes during treatment with olanzapine. BMC Psychiatry. 2010 Sep 14;10:72. doi: 10.1186/1471-244X-10-72. PMID 20840778
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine: olanzapine plus behavioral information. olanzapine: 5-20 milligrams (mg), oral, daily for 22 weeks.
- Olanzapine + Amantadine: Olanzapine and Pharmacological Algorithm 1a - amantadine first plus behavioral information.
  olanzapine: 5-20 milligrams (mg), oral, daily for 22 weeks. amantadine: 100 mg, oral, twice a day. zonisamide: 100-400 mg, oral, daily (only if patient gained greater than 3 kilograms).
- Olanzapine + Metformin: Olanzapine and Pharmacological Algorithm 1b - metformin first plus behavioral information.
  olanzapine: 5-20 milligrams (mg), oral, daily for 22 weeks. metformin: 500 mg, oral, twice a day for 2 weeks, titrated to 500 mg three times a day thereafter. zonisamide: 100-400 mg, oral, daily (only if patient gained greater than 3 kilograms).
Period: Overall Study
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Started | 50 | 76 | 73
Completed | 39 | 50 | 50
Not Completed | 11 | 26 | 23
Not completed — Adverse Event | 2 | 8 | 4
Not completed — Clinical Relapse | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — Physician Decision | 2 | 0 | 1
Not completed — Protocol Violation | 1 | 2 | 3
Not completed — Sponsor Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 12 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin | Total
Number analyzed (Participants) | 50 | 76 | 73 | 199
Age Continuous [Mean (Standard Deviation); unit: years] | 38.7 (12.89) | 38.2 (11.40) | 38.7 (12.01) | 38.5 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 30 | 30 | 79
  Male | 31 | 46 | 43 | 120
Region of Enrollment [Number; unit: participants]
  United States | 13 | 22 | 21 | 56
  Mexico | 7 | 9 | 11 | 27
  Puerto Rico | 5 | 8 | 5 | 18
  Israel | 5 | 8 | 9 | 22
  Russian Federation | 11 | 15 | 14 | 40
  Korea, Republic of | 9 | 14 | 13 | 36
Race/Ethnicity [Number; unit: participants]
  African | 2 | 10 | 4 | 16
  Caucasian | 23 | 30 | 34 | 87
  East Asian | 10 | 15 | 14 | 39
  Hispanic | 14 | 20 | 18 | 52
  Native American | 0 | 0 | 1 | 1
  West Asian | 1 | 1 | 2 | 4
Type of Diagnosis [Number; unit: participants]
  Schizoaffective | 8 | 15 | 18 | 41
  Schizophrenia | 42 | 61 | 55 | 158
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meter (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meter (kg/m^2) | 27.0 (4.53) | 27.3 (4.67) | 27.0 (4.84) | 27.1 (4.68)
Onset Age [Mean (Standard Deviation); unit: years] | 24.35 (8.42) | 26.44 (9.98) | 24.40 (9.18) | 25.15 (9.32)
Previous Number of Episodes [Mean (Standard Deviation); unit: number of episodes] | 1.53 (1.02) | 2.19 (5.90) | 2.22 (5.77) | 2.04 (5.06)
Weight [Mean (Standard Deviation); unit: kilograms] | 77.0 (16.33) | 79.1 (17.27) | 76.2 (16.22) | 77.5 (16.62)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint in Weight
Time Frame: Baseline to endpoint (22 weeks)
Population: All randomized participants with baseline and at least one postbaseline measurement.
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Number analyzed (Participants) | 40 | 50 | 51
kilograms | 2.76 (0.75) | 2.40 (0.65) | 0.65 (0.63)
Statistical Analysis 1: Comparison: Olanzapine vs Olanzapine + Amantadine vs Olanzapine + Metformin; To detect a difference between treatment arms of 3.06 kg in mean weight change from baseline to endpoint, 150 patients must be enrolled in stepped intervention arm and 50 in control arm. Assuming a standard deviation of 6.87 kg, there is 80% power to detect a difference between treatment arms on a 1-sided 2-sample t-test at the 5% significance level. Primary analysis was the comparison of mean weight change for 'olanzapine only' versus pooled 'olanzapine & adjunctive treatment' arm at Week 22; Test type: Superiority or Other; p = 0.065, Mixed Models Analysis — P-value for Olanzapine versus pooled olanzapine+amantadine and olanzapine+metformin; Repeated Measures Analysis
Statistical Analysis 2: Comparison: Olanzapine vs Olanzapine + Amantadine; Hypothesis=weight gain associated with olanzapine can be prevented or mitigated with an adjunctive pharmacological algorithm; Test type: Superiority or Other; p = 0.113, Mixed Models Analysis; Repeated Measures Analysis
Statistical Analysis 3: Comparison: Olanzapine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis; Repeated Measures Analysis

2. Secondary Outcome: Mean Change From Baseline to Endpoint in Fasting Triglycerides
Time Frame: Baseline to endpoint (22 weeks)
Population: All randomized participants with baseline and at least one postbaseline measurement. Last post-baseline measurement carried forward.
Measure: Mean (Standard Deviation); unit: millimoles per Liter (mmol/L)
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Number analyzed (Participants) | 42 | 49 | 56
millimoles per Liter (mmol/L)
  Baseline | 1.58 (0.81) | 1.61 (0.76) | 1.68 (1.00)
  Change from Baseline | 0.33 (1.01) | 0.35 (0.88) | 0.06 (0.64)
Statistical Analysis 1: Comparison: Olanzapine vs Olanzapine + Amantadine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.498, ANCOVA — P-value for Change from Baseline for Olanzapine versus pooled olanzapine+amantadine and olanzapine+metformin
Statistical Analysis 2: Comparison: Olanzapine vs Olanzapine + Amantadine; Test type: Superiority or Other; p = 0.637, ANCOVA — P-value for Change from Baseline
Statistical Analysis 3: Comparison: Olanzapine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.125, ANCOVA — P-value for Change from Baseline

3. Secondary Outcome: Mean Change From Baseline to Endpoint in Fasting Total Cholesterol
Time Frame: Baseline to endpoint (22 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Number analyzed (Participants) | 42 | 49 | 56
millimole per Liter (mmol/L)
  Baseline | 5.01 (1.00) | 5.03 (1.09) | 4.91 (1.21)
  Change from Baseline | 0.36 (0.84) | 0.01 (1.06) | -0.08 (0.92)
Statistical Analysis 1: Comparison: Olanzapine vs Olanzapine + Amantadine; Test type: Superiority or Other; p = 0.173, ANCOVA — P-value for Change from Baseline
Statistical Analysis 2: Comparison: Olanzapine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.016, ANCOVA — P-value for Change from Baseline
Statistical Analysis 3: Comparison: Olanzapine vs Olanzapine + Amantadine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.029, ANCOVA — P-value for Change from Baseline for Olanzapine versus pooled olanzapine+amantadine and olanzapine+metformin

4. Secondary Outcome: Mean Change From Baseline to Endpoint in Fasting High Density Lipoprotein (HDL) Cholesterol
Time Frame: Baseline to endpoint (22 weeks)
Population: Number of randomized participants with a baseline and at least one post-baseline measurement. Last post-baseline measurement carried forward.
Measure: Mean (Standard Deviation); unit: millimole per liter (mmol/L)
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Number analyzed (Participants) | 46 | 63 | 64
millimole per liter (mmol/L)
  Baseline | 1.25 (0.29) | 1.26 (0.36) | 1.22 (0.35)
  Change from Baseline | -0.00 (0.23) | -0.11 (0.25) | -0.08 (0.24)
Statistical Analysis 1: Comparison: Olanzapine vs Olanzapine + Amantadine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.017, ANCOVA — P-value for Change from Baseline for Olanzapine versus pooled olanzapine+amantadine and olanzapine+metformin
Statistical Analysis 2: Comparison: Olanzapine vs Olanzapine + Amantadine; Test type: Superiority or Other; p = 0.015, ANCOVA — P-value for Change from Baseline
Statistical Analysis 3: Comparison: Olanzapine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.071, ANCOVA — P-value for Change from Baseline

5. Secondary Outcome: Mean Change From Baseline to Endpoint in Fasting Low Density Lipoprotein (LDL) Cholesterol
Time Frame: Baseline to endpoint (22 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Number analyzed (Participants) | 40 | 47 | 55
millimole per Liter (mmol/L)
  Baseline | 3.02 (0.88) | 3.06 (1.03) | 2.91 (0.93)
  Change from Baseline | 0.16 (0.60) | -0.04 (0.95) | -0.02 (0.84)
Statistical Analysis 1: Comparison: Olanzapine vs Olanzapine + Amantadine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.152, ANCOVA — P-value for Change from Baseline for Olanzapine versus pooled olanzapine+amantadine and olanzapine+metformin
Statistical Analysis 2: Comparison: Olanzapine vs Olanzapine + Amantadine; Test type: Superiority or Other; p = 0.350, ANCOVA — P-value for Change from Baseline
Statistical Analysis 3: Comparison: Olanzapine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.123, ANCOVA — P-value for Change from Baseline

6. Secondary Outcome: Mean Change From Baseline to Endpoint in Fasting Glucose
Time Frame: Baseline to endpoint (22 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimole per Liter (mmol/L)
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Number analyzed (Participants) | 44 | 59 | 64
millimole per Liter (mmol/L)
  Baseline | 5.32 (0.46) | 5.25 (0.78) | 5.28 (0.63)
  Change from Baseline | 0.26 (0.99) | 0.10 (0.48) | 0.01 (0.58)
Statistical Analysis 1: Comparison: Olanzapine vs Olanzapine + Amantadine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.499, ANCOVA — P-value for Change from Baseline for Olanzapine versus pooled olanzapine+amantadine and olanzapine+metformin
Statistical Analysis 2: Comparison: Olanzapine vs Olanzapine + Amantadine; Test type: Superiority or Other; p = 0.833, ANCOVA — P-value for Change from Baseline
Statistical Analysis 3: Comparison: Olanzapine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.339, ANCOVA — P-value for Change from Baseline

7. Secondary Outcome: Mean Change From Baseline to Endpoint in Hemoglobin A1c
Time Frame: Baseline to endpoint (22 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent hemoglobin A1c
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Number analyzed (Participants) | 44 | 63 | 63
percent hemoglobin A1c
  Baseline | 5.51 (0.46) | 5.48 (0.39) | 5.53 (0.37)
  Change from Baseline | 0.09 (0.45) | 0.10 (0.37) | -0.03 (0.25)
Statistical Analysis 1: Comparison: Olanzapine vs Olanzapine + Amantadine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.278, ANCOVA — P-value for Change from Baseline for Olanzapine versus pooled olanzapine+amantadine and olanzapine+metformin
Statistical Analysis 2: Comparison: Olanzapine vs Olanzapine + Amantadine; Test type: Superiority or Other; p = 0.976, ANCOVA — P-value for Change from Baseline
Statistical Analysis 3: Comparison: Olanzapine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.049, ANCOVA — P-value for Change from Baseline

8. Secondary Outcome: Change From Baseline to Endpoint in Brief Psychiatric Rating Scale (BPRS) Total Score
Description: The BPRS is an 18-item clinician-administered scale used to assess the degree of severity of a subject's general psychopathological symptoms. Each item is rated on a scale from 1 (symptom not present) to 7 (symptom extremely severe). The BPRS total score ranges from 18 to 126.
Time Frame: Baseline to endpoint (22 weeks)
Population: Number of participants with a baseline and at least one post baseline measurement. Last post-baseline measurement carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Number analyzed (Participants) | 45 | 67 | 72
units on a scale
  Baseline | 48.24 (15.98) | 45.90 (12.44) | 47.00 (14.18)
  Change from Baseline | -13.89 (18.61) | -9.90 (11.24) | -9.72 (14.15)
Statistical Analysis 1: Comparison: Olanzapine vs Olanzapine + Amantadine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.122, ANCOVA — P-value for Change from Baseline for Olanzapine versus pooled olanzapine+amantadine and olanzapine+metformin
Statistical Analysis 2: Comparison: Olanzapine vs Olanzapine + Amantadine; Test type: Superiority or Other; p = 0.225, ANCOVA — P-value for Change from Baseline
Statistical Analysis 3: Comparison: Olanzapine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.124, ANCOVA — P-value for Change from Baseline

9. Secondary Outcome: Change From Baseline to Endpoint in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a rating scale for severity of depressive mood symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
Time Frame: Baseline to endpoint (22 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Number analyzed (Participants) | 46 | 67 | 72
units on a scale
  Baseline | 12.76 (8.08) | 14.22 (11.14) | 15.40 (9.21)
  Change from Baseline | -6.39 (8.37) | -4.12 (7.20) | -4.36 (7.47)
Statistical Analysis 1: Comparison: Olanzapine vs Olanzapine + Amantadine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.020, ANCOVA — P-value for Change from Baseline for Olanzapine versus pooled olanzapine+amantadine and olanzapine+metformin
Statistical Analysis 2: Comparison: Olanzapine vs Olanzapine + Amantadine; Test type: Superiority or Other; p = 0.037, ANCOVA — P-value for Change from Baseline
Statistical Analysis 3: Comparison: Olanzapine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.038, ANCOVA — P-value for Change from Baseline

10. Secondary Outcome: Change From Baseline to Endpoint in Clinical Global Impression - Severity Scale (CGI-S)
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
Time Frame: Baseline to endpoint (22 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Number analyzed (Participants) | 47 | 72 | 73
units on a scale
  Baseline | 4.06 (1.24) | 4.03 (1.07) | 4.00 (1.13)
  Change from Baseline | -0.98 (1.13) | -0.72 (1.14) | -0.79 (1.03)
Statistical Analysis 1: Comparison: Olanzapine vs Olanzapine + Amantadine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.474, ANCOVA — P-value for Change from Baseline for Olanzapine versus pooled olanzapine+amantadine and olanzapine+metformin
Statistical Analysis 2: Comparison: Olanzapine vs Olanzapine + Amantadine; Test type: Superiority or Other; p = 0.404, ANCOVA — P-value for Change from Baseline
Statistical Analysis 3: Comparison: Olanzapine vs Olanzapine + Metformin; Test type: Superiority or Other; p = 0.652, ANCOVA — P-value for Change from Baseline

11. Secondary Outcome: Correlations Between Weight Changes and Changes in Eating Inventory (EI) and Food Craving Inventory (FCI) at 2 Weeks and 22 Weeks
Description: To understand the drivers of weight gain as indicated by the correlation between weight changes and changes in the Eating Inventory (EI) and Food Craving Inventory (FCI). The EI is a 51-item inventory that measures dietary restraint, disinhibition, and perceived hunger. The FCI is a 28-item instrument measuring the frequency over the past month of general cravings and cravings for specific types of foods, namely: high fats, sweets, carbohydrates/starches, and fast-food fats. Correlations were computed on the combined treatment groups.
Time Frame: Baseline to endpoint (22 weeks)
Population: N=Pairs of Observations for the combined treatment groups.
Measure: Number; unit: correlation
Groups:
- 2 Weeks; 22 Weeks: Combined treatment groups:
  olanzapine plus behavioral information [olanzapine: 5-20 milligrams (mg), oral, daily for 22 weeks].
  Olanzapine and Pharmacological Algorithm 1a - amantadine first plus behavioral information [olanzapine: 5-20 milligrams (mg), oral, daily for 22 weeks. amantadine: 100 mg, oral, twice a day. zonisamide: 100-400 mg, oral, daily (only if patient gained greater than 3 kilograms)].
  Olanzapine and Pharmacological Algorithm 1b - metformin first plus behavioral information [olanzapine: 5-20 milligrams (mg), oral, daily for 22 weeks. metformin: 500 mg, oral, twice a day for 2 weeks, titrated to 500 mg three times a day thereafter. zonisamide: 100-400 mg, oral, daily (only if patient gained greater than 3 kilograms)].
Arm/Group | 2 Weeks | 22 Weeks
Number analyzed (Participants) | 66 | 41
correlation
  EI: Disinhibition | -0.034 | 0.285
  EI: Cognitive Restraint | -0.273 | -0.038
  EI: Hunger | -0.150 | 0.148
  FCI: Carbohydrates/Starches (N=186, N=141) | 0.013 | -0.064
  FCI: Fast Food Fats (N=188, N=140) | -0.019 | 0.047
  FCI: High Fats (N=186, N=138) | 0.051 | 0.043
  FCI: Sweets (N=187, N=140) | 0.022 | -0.008
  FCI: Total Score (N=184, N=137) | 0.039 | -0.000

ADVERSE EVENTS:
Arm/Group | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Serious Adverse Events (participants affected / at risk) | 5 | 4 | 4
Other Adverse Events (participants affected / at risk) | 26 | 38 | 46
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Chest pain (General disorders) | 0/50 (0) | 0/76 (0) | 1/73 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/50 (0) | 1/76 (1) | 0/73 (0)
Akathisia (Nervous system disorders) | 0/50 (0) | 1/76 (1) | 0/73 (0)
Hallucination (Psychiatric disorders) | 0/50 (0) | 1/76 (1) | 2/73 (2)
Panic attack (Psychiatric disorders) | 0/50 (0) | 1/76 (1) | 0/73 (0)
Psychotic disorder (Psychiatric disorders) | 1/50 (1) | 0/76 (0) | 0/73 (0)
Schizophrenia (Psychiatric disorders) | 3/50 (3) | 0/76 (0) | 0/73 (0)
Suicidal ideation (Psychiatric disorders) | 1/50 (1) | 0/76 (0) | 0/73 (0)
Suicide attempt (Psychiatric disorders) | 0/50 (0) | 0/76 (0) | 1/73 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Olanzapine | Olanzapine + Amantadine | Olanzapine + Metformin
Constipation (Gastrointestinal disorders) | 0/50 (0) | 3/76 (3) | 3/73 (3)
Diarrhoea (Gastrointestinal disorders) | 0/50 (0) | 3/76 (3) | 10/73 (11)
Dry mouth (Gastrointestinal disorders) | 2/50 (2) | 4/76 (4) | 0/73 (0)
Nausea (Gastrointestinal disorders) | 2/50 (2) | 3/76 (3) | 5/73 (6)
Vomiting (Gastrointestinal disorders) | 0/50 (0) | 1/76 (1) | 5/73 (5)
Asthenia (General disorders) | 1/50 (1) | 0/76 (0) | 3/73 (3)
Fatigue (General disorders) | 1/50 (1) | 2/76 (2) | 3/73 (3)
Nasopharyngitis (Infections and infestations) | 0/50 (0) | 4/76 (4) | 0/73 (0)
Urinary tract infection (Infections and infestations) | 2/50 (2) | 0/76 (0) | 0/73 (0)
Overdose (Injury, poisoning and procedural complications) | 2/50 (2) | 0/76 (0) | 0/73 (0)
Weight increased (Investigations) | 2/50 (3) | 4/76 (4) | 4/73 (4)
Increased appetite (Metabolism and nutrition disorders) | 3/50 (4) | 1/76 (1) | 3/73 (3)
Akathisia (Nervous system disorders) | 2/50 (2) | 3/76 (3) | 2/73 (2)
Dizziness (Nervous system disorders) | 2/50 (2) | 1/76 (1) | 2/73 (2)
Headache (Nervous system disorders) | 2/50 (2) | 2/76 (2) | 4/73 (4)
Sedation (Nervous system disorders) | 0/50 (0) | 4/76 (4) | 2/73 (2)
Somnolence (Nervous system disorders) | 4/50 (4) | 5/76 (5) | 8/73 (10)
Anxiety (Psychiatric disorders) | 2/50 (2) | 3/76 (3) | 2/73 (2)
Insomnia (Psychiatric disorders) | 5/50 (5) | 4/76 (5) | 1/73 (3)
Sleep disorder (Psychiatric disorders) | 2/50 (2) | 0/76 (0) | 1/73 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days